CLINICAL TRIAL: NCT06899607
Title: Bridging the Fibre Gap: A Pre-post Single-arm Feasibility Trial on Increased Fibre Intake and Mental Wellbeing
Brief Title: Fibre and Mental Wellbeing Feasibility Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Responsible Party: Principal Investigator, Piril Hepsomali, Principle Investigator, University of Reading
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2025-037-PH
Record Dates: First submitted 2025-03-25; First posted 2025-03-28 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Affect (Mental Function); Sleep; Anxiety; Stress
Keywords: fibre; depression; anxiety; stress; optimism; sleep; gut health
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fibre arm (Experimental)
  Interventions: Other: Fibre arm

INTERVENTIONS:
Other: Fibre arm — Increasing daily fibre intake by 10 grams

SUMMARY:
This feasibility study will explore whether adding an extra 10 grams of fibre to participants' daily diet for two weeks would improve their mental health and wellbeing.

DETAILED DESCRIPTION:
The current pre-post single-arm feasibility trial will investigate whether increasing daily fibre intake by 10 grams for two weeks enhance depression, anxiety, stress, sleep quality, gut health, and optimism in 18-40 year-old young adults. Participants will be provided a list of high fibre food items. Outcome measures will be acquired before and after 2-weeks . These will include cognitive measures of measures of depression, anxiety, and stress symptomatology; sleep; gastrointestinal symptomatology; optimism.

ELIGIBILITY:
Inclusion Criteria:

* Aging between 18-40 years old
* Having normal vision and hearing
* Having a body mass index between 18.5 and 30
* Not following a high fibre diet >20g fibre/day as assessed by using the FiberScreen

Exclusion Criteria:

* Smoking
* Having food allergies
* Following restrictive and/or unbalanced diets
* Changing dietary intake majorly in past month
* Being diagnosed with any psychiatric or neurologic conditions
* Being diagnosed with any cardiometabolic diseases, or hypertension or thrombosis related disorders or suffer from thyroid disease
* Currently taking anticoagulants, antiplatelet medication, antidepressants, proton-pump inhibitors
* Currently consuming prebiotic or probiotic supplements or laxatives
* Continuous antibiotic use for > 3 days within 1 month prior to enrolment
* Continuous use of weight-loss drug for > 1 month before screening
* Having a significant gastrointestinal (GI) condition

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2027-09-05 (Estimated); Study Completion 2027-09-05 (Estimated)

PRIMARY OUTCOMES:
Generalized Anxiety Disorder 7 scale scores | From baseline (pre intervention) to week 2 (post intervention)
  A validated self-report measure of anxiety
Patient Health Questionaire-8 scores | From baseline (pre intervention) to week 2 (post intervention)
  A validated self-report measure of depression
Perceived Stress Scale scores | From baseline (pre intervention) to week 2 (post intervention)
  A validated self-report measure of stress

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index scores | From baseline (pre intervention) to week 2 (post intervention)
  A validated self-report measure of sleep quality
Gastrointestinal Symptom Rating Scale Scores | From baseline (pre intervention) to week 2 (post intervention)
  A validated self-report measure of gastrointestinal symptoms that includes 15-items (combined into five symptom clusters depicting Reflux, Abdominal pain, Indigestion, Diarrhoea and Constipation)
Revised Life Orientation Test Scores | From baseline (pre intervention) to week 2 (post intervention)
  A validated self-report measure of one's dispositional level of optimism

OTHER OUTCOMES:
EPIC Norfolk Food Frequency Questionnaire (FFQ) | Baseline (pre intervention) only
  The FFQ is a validated tool for gauging the average habitual dietary intake of micro and macronutrients of an individual in the UK. Data will be processed using the FETA software.
FiberScreen Scores | From baseline (pre intervention) to week 2 (post intervention)
  A questionnaire that assesses fibre intake. It will be used to screen participants. Individuals who adhere to a high fibre diet (>20g fibre/day) will be excluded from the study.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, School of Psychology and Clinical Languages, Reading, Berkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No